CLINICAL TRIAL: NCT02314910
Title: Exploring Bone Innervation Around Osseointegrated Implants
Brief Title: Bone Innervation Around Implants
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: BAI_040413
Record Dates: First submitted 2013-04-05; First posted 2014-12-11 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Innervation of Bone Around Implants
Keywords: Innervation; Jaw Bone; Implants; Stereognostic; Osseoperception

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Implant surrounded by bone material
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Failed implant: There is only one group, being the group of patients of which the oral implant needed to be removed for clinical reasons.
  Interventions: Other: Sample histology

INTERVENTIONS:
Other: Sample histology

SUMMARY:
If implants are osseointegrated, there might be innervation of the bone close to the implants. This event might explain the so-called osseoperception phenomena: Functioning with implant-supported oral prostheses is better than with removable prostheses due to physiologic integration and thus sensory feedback.

DETAILED DESCRIPTION:
Several studies confirm improved oral functions in patients who wear dentures on implants, compared with patients with a removable denture. This could possibly be explained by sensory innervation around the implant. However, the mechanism of the phenomenon is not yet completely elucidated.

A first step is to identify and describe nerve fibers around implants that are integrated in human jawbone. The results of this study can then be used to identify the factors that promote such innervation (implant surface, surgical procedure, patient-related factors, ...).

Goal The purpose of this study is to identify and characterize nerve fibers around osseogeïntegreerde implants.

Materials and methods Inclusion and exclusion Only implants that were lost due to mechanical failure or because of severe bone loss will be used. In the case of bone loss, an analysis will only be performed if sufficient osseointegration took place apical to the implant, at least about ¼ of the length of the implant. All these failed implants should be removed from a clinical point of view, but the extensive osseointegration purpose necessitates the clinical use of a trepanbur, a cylindrical bur to remove jaw bone. All patients will, prior to surgery, give informed consent to use their implants for further research, as well as the data from their clinical file.

Collection of samples It is not possible to identify nerve fibers around the implants on the basis of radiological images, because the resolution is not high enough and because radiology of material with very high density (titanium) results in a distorted picture, exactly in the space around the implant . Therefore, a histological analysis will be made on the implants.

For this study, over a period of 5 years, as far as possible, implants will be collected with a minimum of 20. The implants will be collected from patients in three clinical centers where implants are placed: UZ Leuven, ZOL Genk and a private practice in Leuven.

The implants are removed with a trepanbur and immediately preserved in glutaraldehyde or formaldehyde.

Analysis of the samples The fixed samples are decalcified in 10% EDTA, hydrated through graded concentrations of ethanol and finally placed in Araldite. They can then be cut with a bonemicrotome (Reichert Ultracut E Microtome, Vienna, Austria) and further prepared for light microscopic and ultrastructural analysis. Staining with methylene blue (0.1% aqueous solution) will be done on sections of 0.5 um. These sections will be viewed with a light microscope and digitized at a high resolution Mirax Scan (Carl Zeiss Micro-Imaging GmbH, Germany). The images will be evaluated by an expert at a magnification of 20x, 40x and 100x on a 30inch LCD screen with custom software (Mirax Viewer 1.1, Göttingen, Germany). For the analysis of the ultrastructural features, the investigators will make ultrathin sections (0.06μm) and on plates coated with 0.7% formvar places, contrasted with uranyl acetate and lead citrate. These sections are EM208S analyzed with a transmission electron microscope (Philips, Eindhoven, The Netherlands) at 80 kV.

Expected results Following a pilot study, the investigators expect in certain cases to discover new nerve fibers in bone around implants. These nerve fibers can be described, and their nature identified. If sufficient fibers are detected with these results, the investigators can prove the osseoperception phenomena. This information can then be used for the optimization of therapies with implants, so that the best possible integration, both biologically and physiologically, can take place.

ELIGIBILITY:
Inclusion Criteria:

* Implant lost due to clinical reasons

Exclusion Criteria:

* No osseointegration

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients of which the implant needed to be removed
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-08; Primary Completion 2018-07 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Nerve fibre detection | 1 year
  To detect a newly formed nerve fibre close to the implant

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium